CLINICAL TRIAL: NCT05245318
Title: Cost-effectiveness of a Smartphone Application for Tinnitus Treatment (The CATT Trial): A Study Protocol of a Randomised Controlled Trial
Brief Title: The CATT Trial: Cost-effectiveness of a Smartphone Application for Tinnitus Treatment
Acronym: CATT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Universiteit Antwerpen (Other); University Hospital, Antwerp (Other); University of Regensburg (Other)
Responsible Party: Principal Investigator, Sarah Michiels, Prof. Dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T002221N
Record Dates: First submitted 2022-01-26; First posted 2022-02-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Tinnitus
Keywords: somatic tinnitus; smartphone application; telerehabilitation; blended physiotherapy program
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-blind two-arm 1:1 randomised controlled trial. The study is designed as a non-inferiority trial of a continuous response variable comparing independent control and experimental subjects. After baseline measurements, patients will be randomised into either the experimental group or the control group. A stratified randomisation according to the grade of tinnitus severity obtained by use of the Tinnitus Functional Index (TFI) and gender will be used. A minimisation procedure will be used to perform the stratified randomisation using the web-based online randomisation tool Qminim.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study patients will be blinded towards the group they will be randomised to, but the therapist cannot be blinded, as she knows whether a patient receives the treatment every week or every two weeks. To limit the risk of bias related to lack of blinding of the therapist, all evaluation measurements will be performed by a blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard clinical care control group (Active Comparator): Standard physiotherapy program of 12 weeks (1 treatment session /week)
  Interventions: Other: Standard Clinical care
- Experimental blended physiotherapy program group (Experimental): Blended physiotherapy program of 12 weeks with exercises and counselling provided through a smartphone application and 6 face-to-face treatment sessions (1 physiotherapy treatment session every 2 weeks)
  Interventions: Device: Blended physiotherapy program

INTERVENTIONS:
Other: Standard Clinical care — The standard care treatment comprises 12 face-to-face individual physiotherapy sessions at a ratio of 1 session a week. Every patient in the control group will be treated in a tailored manner according to their results on the baseline measurements. The multimodal treatment program will consist of exercises to increase strength, endurance and coordination of the cervical spine and shoulder stabilising muscles, exercises to increase mobility and improve posture. In case of jaw complaints stretching exercises of the masticatory muscles are added to the program. In addition, manual mobilisations and manual techniques to decrease muscle tension in neck and jaw muscles can be added to the exercise program if necessary. Patients will receive counselling to learn about their neck/jaw complaints but no tinnitus counselling. Patients will be motivated to perform the exercise program at home on a daily basis. Patients will be evaluated weekly.
  Arms: Standard clinical care control group
Device: Blended physiotherapy program — The experimental group will receive a blended physiotherapy program consisting of six physiotherapy treatments over a period of 12 weeks, meaning one treatment session every two weeks. In addition, a smartphone application will offer the patients a daily exercise program, based upon the standard physiotherapy treatment, and psychological counselling. Before the start of the program, the exercises will be tailored to the area, type and degree of the patient's dysfunctions. During the six physiotherapy treatment sessions patients will (if needed), receive additional manual mobilisations to increase mobility of the neck and/or temporomandibular joints or manual techniques to decrease muscle tension in neck and jaw muscles. Additional counselling on knowledge about neck and jaw pain and advice about good posture and movement habits will also be provided by the physiotherapist during these six treatment sessions.
  Arms: Experimental blended physiotherapy program group

SUMMARY:
The twofold aim of this single-blind two-arm 1:1 randomised control trial is to examine if the treatment effect and cost-effectiveness of a smartphone application, designed to increase therapy compliance and provide tinnitus counselling, as part of a blended physiotherapy program, is, as hypothesised, as good as or better in comparison to standard clinical care.

DETAILED DESCRIPTION:
Background: Tinnitus is a highly prevalent symptom with a variety of possible underlying diseases, affecting 10-15% of the adult population. Apart from the heterogenous clinical origin, it is also characterised by a diverse clinical representation, often causing distress and interfering with daily functioning and quality of life. In case the tinnitus is influenced by alterations in somatosensory afference from the cervical spine or temporomandibular area, due to increased muscle tension or movement restrictions, it is referred to as somatic or somatosensory tinnitus (ST). ST is known to react well to physiotherapy treatment, but currently, it is hard to motivate patients to do their home exercises properly and the necessary tinnitus counselling is often lacking.

Objective: The twofold aim of this study is to examine if the treatment effect and cost-effectiveness of a smartphone application, designed to increase therapy compliance and provide tinnitus counselling, as part of a blended physiotherapy program, is, as hypothesised, as good as or better in comparison to standard clinical care.

Methods and design: This study is designed as a single-blind two-arm 1:1 randomised control trial. Adult patients diagnosed with ST, without psychiatric comorbidities and with basic knowledge of the use of a smartphone, will be recruited at the Ear Nose Throat (ENT) department of the Antwerp university hospital (UZA). After inclusion and baseline measurements, patients will be randomised to one of the treatment groups. The experimental group will receive the blended physiotherapy program containing six in-clinic physiotherapy sessions over a period of twelve weeks (1x/2weeks) and access to the exercise and counselling program provided by the smartphone application. The control group will receive the standard care physiotherapy program comprising twelve weekly in-clinic physiotherapy sessions. As a primary outcome measure, the change in Tinnitus Functional Index (TFI) score at 1 month after the last treatment will be used. Secondary outcome measures are the visual analogue scale (VAS) for tinnitus loudness, Neck Bournemouth Questionnaire (NBQ), Temporomandibular disorder (TMD) pain screener, clinical neck and jaw tests, pure tone audiometry, speech-in-quiet (SPIQ) and speech-in-noise (SPIN) understanding, psychoacoustic tinnitus measures (tinnitus pitch and loudness matching), the Hospital Anxiety and Depression Scale (HADS), the Hyperacusis Questionnaire (HQ). Additionally, a cost-effectiveness analysis will be performed informing on both medical costs and indirect costs. Data from the Euroqol EQ-5D and iMTA Productivity Cost Questionnaire (PCQ) will be used in this analysis. Data for all outcome measures will be collected at baseline, one month after the last treatment session and three months after the last treatment session.

Discussion: This is the first study to combine both tinnitus counselling and neck/jaw pain treatment provided by a digital application in a blended physiotherapy program. This is in order to empower ST patients to improve and better manage their own health and possibly reduce economic costs by alleviating the tinnitus burden ST patients experience. The advantages of this single-blind two-arm randomised controlled trial are the high-quality methodological design, the great sample size and the expertise of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Adults (+ 18 years old) with Somatic tinnitus (ST), diagnosed according to the diagnostic criteria for ST
* Fluent in Dutch
* Own smartphone and able to use common applications without support

Exclusion Criteria:

* Other types of tinnitus
* Active middle ear pathology
* An active psychiatric disorder (such as anxiety disorder or clinical depression) diagnosed by the psychiatric team of Antwerp University Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index (TFI) | from baseline to one month follow-up (also tested after last treatment session and at three months follow-up)
  The primary outcome is the change in Tinnitus functional index (TFI) score from baseline to one month after the treatment. This timepoint was chosen since previous research indicated that the largest treatment effect on TFI is to be expected four to seven weeks after the last treatment session. The TFI is a self-report questionnaire comprising 25 questions, each scored by an eleven-point Likert scale, objectifying the impact and severity of tinnitus. Eight subscores are differentiated, namely intrusiveness, sense of control, cognitive complaints, sleep disturbance, auditory difficulties, relaxation, quality of life (QOL) and emotional distress. The total score and subscores are noted on a scale of 0 to 100. Higher scores indicate higher levels of tinnitus-related distress. TFI has a good test-retest reliability (r: 0.78), discriminant validity with the Beck Depression Inventory-Primary Care (r: 0.56) and convergent validity with the Tinnitus Handicap Inventory (THI) (r: 0.86).

SECONDARY OUTCOMES:
Cervical spine mobility | from baseline to one and three months follow-up
  Cervical spine mobility will be measured in degrees using the NeckCare Unit. This device, using accelerometer and gyroscope data, is specifically designed for investigating the cervical range of motion and provides a separate figure for the range of motion in each movement plane.
Joint Repositioning Accuracy (JRA) | from baseline to one and three months follow-up
  Joint repositioning accuracy (JRA) after flexion, extension and left and right rotation movements will be measured in degrees using the NeckCare Unit. This device, using accelerometer and gyroscope data, is specifically designed for investigating JRA during head-neck relocation tests.
Strength of deep neck flexors | from baseline to one and three months follow-up
  The strength of the deep neck flexor muscles will be assessed according to the standardized protocol proposed by Segarra et al.. The patient lays down in supine position and is asked to lift the head of the table, while holding a double chin. This test is graded by the amount of seconds that the patient can hold this position correctly.
Coordination of deep neck extensors | from baseline to one and three months follow-up
  The coordination of the deep neck extensor muscles will be assessed according to the standardized protocol proposed by Segarra et al..he deep neck extensor test will be performed in a four-point-kneeling position. The test will be assessed based on the fulfilment of certain criteria such as presence of dissociation between mid-low cervical and high cervical spine, neutral head position during 20° mid-low cervical extension, absence poked chin, absence excessive tension of Musculus Semispinalis Capitis.
Coordination of shoulder stabilizing muscles | from baseline to one and three months follow-up
  The coordination of the shoulder stabilising muscles will be assessed according to the standardized protocol proposed by Segarra et al.. The scapula stabilisation test will be performed in prone position with one arm elevated. The patient should perform a shoulder depression and lift the elevated arm, without losing the shoulder depression. In case a patient can perform the test correctly, he will be scored as good coordination. All other cases will be scored as bad coordination.
Jaw mobility | from baseline to one and three months follow-up
  The mobility of the temporomandibular joint will be measured using a ruler. Mouth opening, protrusion and laterotrusion will be objectified.
Myofascial triggerpoints | from baseline to one and three months follow-up
  Active myofascial trigger points will be looked for in the masseter and temporalis muscle and in the sternocleidomastoid, splenius capitis, upper trapezius and levator scapulae muscles. A triggerpoint is considered active when a patient indicated that pressure on the triggerpoint was painful not only locally but also in the radiation area of the respective trigger point.
Pure tone hearing thresholds | from baseline to one and three months follow-up
  Pure tone audiometry, to objectify the presence of hearing loss, is performed according to current clinical standards (ISO 8253-1, 1989) using a two-channel Interacoustics AC-40 audiometer in a silent room. Air conduction thresholds are measured by the use of headphones at 125Hz, 250Hz, 500Hz, 1 kHz, 2 kHz, 3 kHz, 4 kHz, 6 kHz and 8 kHz. In cases where air conduction thresholds exceed the normality level of 20dB HL at one frequency between 250Hz and 4 kHz, bone conduction thresholds are measured.
Speech-in-quiet (SPIQ) understanding | from baseline to one and three months follow-up
  Speech reception in quiet (SPIQ) is measured using the Dutch open-set NVA lists developed by the Nederlandse Vereniging voor Audiologie (NVA) or Dutch Society for Audiology. Each list consists of twelve monosyllabic words (consonant-vowel-consonant), of which one is a training item. The speech recognition score is the percentage of correctly identified phonemes. The lists are presented through headphones. The speech reception in noise
Speech-in-noise (SPIN) understanding | from baseline to one and three months follow-up
  The speech reception in noise (SPIN) is assessed by means of the Leuven Intelligibility Sentences Test (LIST) using an adaptive procedure. The frequency spectrum of the noise signal is equal to the long-term average speech spectrum of the sentences. The level of the noise is fixed at 65 dB SPL, while the level of the speech signal is altered depending on the response of the patient. If the participant repeats the keywords of the sentence correctly, the level of the next sentence is decreased by 2 dB SPL. If the participant fails to repeat the keywords, the level is increased
Tinnitus pitch matching | from baseline to one and three months follow-up
  The pitch is the psychoacoustic equivalent of the physical parameter frequency. The tinnitus pitch is obtained by use of a pitch matching technique which is the quantitative and qualitative description of the spectral characteristics of the tinnitus. For this technique, a two-alternative forced-choice procedure was used using the contralateral ear as the reference ear. In cases where tinnitus is perceived bilaterally, the choice of the ear is arbitrary. By this technique, an attempt is made to identify the centre pitch of the tinnitus. When multiple tinnitus sounds are perceived, it is suggested to concentrate on the most troublesome tinnitus sound. Each time a pair of pure tones (or noises in case of noise-like tinnitus), differing by one or more octaves, are presented to the subject, who has to indicate which of the tones resembles the tinnitus the most. This procedure is repeated, and finer adjustments are made to obtain a match of tinnitus pitch as exact as possible.
Tinnitus Loudness matching | from baseline to one and three months follow-up
  Loudness is the perceptual correlate of the sound intensity. The tone (or noise) defined as the pitch math is presented to the ipsilateral ear (when appropriate), and a loudness match is made by the use of an alternating forced-choice procedure.
VAS for tinnitus loudness | from baseline to one and three months follow-up
  Patients are asked to score the mean and maximum loudness of their tinnitus in the previous week on a 100 mm horizontal line ranging from left: 0 (absence of tinnitus) to right: 100 (as loud as possible, cannot be any louder).
Neck Bournemouth Questionnaire (NBQ) score | from baseline to one and three months follow-up
  The presence and severity of neck complaints will be evaluated using the NBQ. The NBQ consists of seven questions on the severity of the neck complaints and its interference with the patient's wellbeing and professional and daily activities. The test-retest reliability of the NBQ is moderate (ICC: 0.65). The construct validity is acceptable with both the Neck Disability Index (r: 0.50) and the Copenhagen Neck Functional Index (r: 0.44). The effect size was high (Cohen's d: 1.67), which indicates that the NBQ is highly responsive to changes in cervical spine complaints. The clinically relevant change of the NBQ is a 12 points decrease.
Temporomandibular disorder (TMD) pain screener score | from baseline to one and three months follow-up
  The presence and severity of temporomandibular disorders (TMD) will be evaluated using the TMD pain screener. The TMD pain screener is a 6-item questionnaire regarding pain complaints from the orofacial region, and their dependency on functions, like opening wide or chewing. Internal consistency of the questionnaire is excellent, with a coefficient α value of 0.93, reliability is good (ICC: 0.79), and excellent sensitivity and specificity for diagnosing TMD (0.99 and 0.95-0.98, respectively).
Hospital Anxiety and Depression Scale (HADS) | from baseline to one and three months follow-up
  The Hospital Anxiety and Depression Scale (HADS) is used to detect signs of depression and anxiety symptoms. It is a self-assessment scale and was developed to identify the possibility and probability of the presence of anxiety and depression among patients in non-psychiatric clinics. It exists of two subscales, an anxiety subscale (HADS-A) and a depression subscale (HADS-D), both containing seven intermingled items. A high internal consistency was stated for a both the depression and anxiety scale, with respectively a mean coefficient α value of 0.83 and 0.82 . In addition both scales also demonstrated a good sensitivity and specificity of approximately 0.80. The HADS is found to be an instrument of moderate reliability (ICC: 0.56) for screening states of depression and anxiety in the setting of a hospital medical outpatient clinic.
Hyperacusis Questionnaire (HQ) | from baseline to one and three months follow-up
  Hyperacusis, a symptom that often co-occurs with tinnitus, is quantified and characterised using the Dutch version of the Hyperacusis Questionnaire (HQ). This questionnaire consists of 14 questions that are answered on a 4-point scale, ranging from 'No' (0 points), 'Yes, a little' (1 point), 'Yes, quite a lot' (2 points) to 'Yes, a lot' (3 points). Scores on the HQ consequently range from 0 to 42, and the cut-off value for hyperacusis is 28 points. Moderate correlations between the HQ, uncomfortable loudness levels, and other health questionnaires and a high Internal consistency of the HQ have been demonstrated.
EuroQol (EQ-5D) | baseline, after last treatment session and at one and three months follow-up
  The EuroQoL EQ-5D questionnaire is the most commonly used method to collect health-related Quality of Life (QoL) data and is recommended by worldwide economic evaluation guidelines such as the NICE recommendations. This questionnaire measures QoL using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The response pattern produces a code which represents a health state of the participant. Each health state is associated with a health utility value between 0 and 1 in which 0 represents death and 1 corresponds to perfect health. QoL is necessary to calculate Quality-Adjusted Life Years (QALYs), the most important outcome from the health economics point of view. The 5L-version is preferred over the 3L-version as it is more nuanced and thus more sensitive to gains (or losses) in general health.
Productivity Cost Questionnaire (iPCQ) | monthly between baseline and three months follow-up
  The iMTA Productivity Cost Questionnaire (iPCQ) includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism (productivity loss due to paid work) and productivity losses related to 3) unpaid work. The iPCQ delivers the necessary input to calculate productivity loss using the Human Capital Approach in the extended analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Demoen S, Jacquemin L, Timmermans A, Van Rompaey V, Vanderveken O, Vermeersch H, Joossen I, Van Eetvelde J, Schlee W, Marneffe W, Luyten J, Gilles A, Michiels S. Cost-effectiveness of a smartphone Application for Tinnitus Treatment (the CATT trial): a study protocol of a randomised controlled trial. Trials. 2022 May 23;23(1):435. doi: 10.1186/s13063-022-06378-7. PMID 35606823